CLINICAL TRIAL: NCT00303043
Title: Hemodynamic Monitoring. The Continuous Measurement of Mixed Venous Saturation Compared to Clinical Valuation: A Pilot Study
Brief Title: Hemodynamic Monitoring With Mixed Venous Saturation
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Davide Chiumello, Policlinico Hospital
Other Study IDs: 2000
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2009-03

CONDITIONS: Critically Ill
Keywords: Hemodynamic monitoring; Mixed venous saturation; Critically ill patients
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: Mixed venous saturation monitoring

INTERVENTIONS:
Procedure: Mixed venous saturation monitoring — Mixed venous saturation monitoring

SUMMARY:
In this study the investigators aim to evaluate the utility of a continuous mixed venous saturation monitoring compared to a clinical examination in a group of critically ill patients.

DETAILED DESCRIPTION:
We will compare possible difference in terms of sensibility and specificity regarding the continuous mixed venous saturation monitoring compared to clinical examination in a group of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients with a central venous catheter

Exclusion criteria:

* Patients with pulmonary catheter

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients with a central venous catheter
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Fondazione Ospedale Maggiore Policlinico Mangiagalli Regina Elena
Locations (1):
- Fondazione Ospedale Maggiore Policlinico Mangiagalli Regina Elena, Milan, mi, Italy